CLINICAL TRIAL: NCT00733265
Title: Study to Investigate the Effects of AZD6140 in Patients With Renal Impairment and in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Jay Horrow, MD, Medical Science Director, AZD6140, AstraZeneca Pharmaceuticals
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D5130C00015; AZD6140/Renal Study
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Renal Impairment
Keywords: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD6140 (Experimental)
  Interventions: Drug: AZD6140

INTERVENTIONS:
Drug: AZD6140 — single oral dose

SUMMARY:
The main purpose of this study is to examine how AZD6140 affects patients with severe kidney disease compared to volunteers with normal kidneys. Subjects in the study will receive one dose of AZD6140.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have severe kidney disease
* Subjects who are matched to the kidney disease patients in terms of weight, age, and sex must have normal kidneys
* All women must be post-menopausal (no longer menstruating) or surgically sterile

Exclusion Criteria:

* Patients requiring dialysis
* History of allergy to aspirin or clopidogrel
* Have increased bleeding risk (for instance uncontrolled high blood pressure or a recent major injury)
* Recent history of fainting or light-headedness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Blood levels of AZD6140 in patients with severe kidney disease compared to volunteers with normal kidneys | Scheduled times during the 3 days after the study drug is taken

SECONDARY OUTCOMES:
Safety and tolerability of AZD6140 in patients with severe kidney disease compared to subjects with normal kidneys | Screening through completion of the study
Measure the effect of AZD6140 on how well blood clots in patients with severe kidney disease compared to subjects with normal kidneys | Scheduled times during the 3 days after the study drug is taken

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Butler, MD, Study Director — AstraZeneca
Locations (4):
- United States (4):
  - Research Site, Phoenix, Arizona
  - Research Site, Anaheim, California
  - Research Site, Miami, Florida
  - Research Site, San Antonio, Texas

REFERENCES:
- [Derived] Butler K, Teng R. Pharmacokinetics, pharmacodynamics, and safety of ticagrelor in volunteers with severe renal impairment. J Clin Pharmacol. 2012 Sep;52(9):1388-98. doi: 10.1177/0091270011415526. Epub 2011 Sep 29. PMID 21960668